CLINICAL TRIAL: NCT02938494
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Study to Compare the Safety and Efficacy of IDP-123 Lotion to Tazorac® (Tazarotene) Cream, in the Treatment of Acne Vulgaris
Brief Title: Safety and Efficacy of IDP-123 Lotion to Tazorac® Cream, in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-123A-201
Record Dates: First submitted 2016-10-11; First posted 2016-10-19 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDP-123 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-123 Lotion
- Tazorac Cream (Active Comparator): Cream
  Interventions: Drug: Tazorac Cream
- Vehicle Lotion (Active Comparator): Lotion
  Interventions: Drug: Vehicle Lotion
- Vehicle Cream (Active Comparator): Cream
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: IDP-123 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-123 Lotion
Drug: Tazorac Cream — Cream
  Other Names: Tazorac
  Arms: Tazorac Cream
Drug: Vehicle Lotion — Lotion
  Other Names: Vehicle
  Arms: Vehicle Lotion
Drug: Vehicle Cream — Cream
  Other Names: Vehicle
  Arms: Vehicle Cream

SUMMARY:
Safety and Efficacy of IDP-123 Lotion (0.045% tazarotene) to Tazorac® (tazarotene) Cream, 0.1%, in the Treatment of Acne Vulgaris

DETAILED DESCRIPTION:
A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Study to Compare the Safety and Efficacy of IDP-123 Lotion (0.045% tazarotene) to Tazorac® (tazarotene) Cream, 0.1%, in the Treatment of Acne Vulgaris

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at least 12 years of age and older.
* Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit).
* Women of childbearing potential and females that are pre-menses must be willing to practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months, IUD, condom with spermicidal, diaphragm with spermicidal, implant, Nuvaring, injection, transdermal patch or abstinence.) Females on birth control pills must have taken the same type pill for at least three months prior to entering the study and must not change type during the study. Those who have used birth control pills in the past must have discontinued usage at least three months prior to the start of the study. Women who use birth control for acne control only should be excluded.
* Pre-menses females and women of childbearing potential must have a negative urine pregnancy test at the screening and baseline visits.

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study;
* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gramnegative folliculitis, dermatitis, eczema.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Subjects with a facial beard or mustache that could interfere with the study assessments.
* Evidence or history of cosmetic-related acne.
* Subject has a history of experiencing significant burning or stinging when applying any facial treatment (eg, make-up, soap, masks, washes, sunscreens, etc) to their face.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (16):
- United States (16):
  - Valeant Site 03, Encinitas, California
  - Valeant Site 04, Fremont, California
  - Valeant Site 06, Los Angeles, California
  - Valeant Site 14, Sacramento, California
  - Valeant Site 01, Santa Monica, California
  - Valeant Site 05, Colorado Springs, Colorado
  - Valeant Site 08, Coral Gables, Florida
  - Valeant Site 10, Miami, Florida
  - Valeant Site 09, Miramar, Florida
  - Valeant Site 12, Louisville, Kentucky
  - Valeant Site 13, Louisville, Kentucky
  - Valeant Site 02, Rockville, Maryland
  - Valeant Site 07, Fridley, Minnesota
  - Valeant Site 16, Chapel Hill, North Carolina
  - Valeant Site 15, High Point, North Carolina
  - Valeant Site 11, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-123 Lotion | Tazorac Cream | Vehicle Lotion | Vehicle Cream
Started | 69 | 72 | 34 | 35
Completed | 65 | 63 | 30 | 31
Not Completed | 4 | 9 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-123 Lotion | Tazorac Cream | Vehicle Lotion | Vehicle Cream | Total
Number analyzed (Participants) | 69 | 72 | 34 | 35 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (10.2) | 22.0 (8.96) | 21.2 (9.27) | 21.2 (7.96) | 22.2 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 17 | 21 | 116
  Male | 32 | 31 | 17 | 14 | 94

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Mean Noninflammatory Lesion Count to Week 12
Description: Noninflammatory lesions were defined as follows: Open comedones (blackhead) - plugged hair follicle with dilated/open orifice, black in color; and Closed comedones (whitehead) - plugged hair follicle: small opening at skin surface. For noninflammatory facial lesions, open and closed comedones were recorded as a single count.
Time Frame: Baseline (Day 0), Week 12
Population: Efficacy analyses compared IDP-123 Lotion and the combined Vehicle Lotion and Vehicle Cream groups, as pre-specified in the statistical analysis plan. There is no information for separate Vehicle Lotion and Vehicle Cream groups, since the comparator group was pre-specified to be combined Vehicle Lotion and Vehicle Cream.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- IDP-123 Lotion: 0.045% tazarotene
- Tazorac Cream: Tazorac Cream 0.1%
- Vehicle Lotion and Vehicle Cream Combined: Vehicle Lotion and Vehicle Cream Combined
Arm/Group | IDP-123 Lotion | Tazorac Cream | Vehicle Lotion and Vehicle Cream Combined
Number analyzed (Participants) | 69 | 72 | 69
lesions | -21.6 (13.98) | -20.3 (13.67) | -13.1 (13.62)

2. Primary Outcome: Absolute Change From Baseline in Mean Inflammatory Lesion Count to Week 12
Description: Inflammatory lesions were defined as follows: Papule - a solid, elevated lesion less than 5 millimeters (mm); and Pustule - an elevated lesion containing pus less than 5 mm. For inflammatory facial lesions, papules and pustules were recorded as a single count, while nodular lesions were counted and recorded separately.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | IDP-123 Lotion | Tazorac Cream | Vehicle Lotion and Vehicle Cream Combined
Number analyzed (Participants) | 69 | 72 | 69
lesions | -18.1 (8.99) | -16.8 (10.96) | -14.0 (8.64)

3. Primary Outcome: Percentage of Participants With Treatment Success at Week 12
Description: Treatment success was defined as at least a 2-grade reduction from Baseline in EGSS score and an EGSS score equating to "Clear" or "Almost Clear". EGSS was based on a 5-point scale ranging from 0 to 4; where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IDP-123 Lotion | Tazorac Cream | Vehicle Lotion and Vehicle Cream Combined
Number analyzed (Participants) | 69 | 72 | 69
Participants | 13 | 12 | 7

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Randomized participants who used study drug at least once and provided ≥1 post-Baseline evaluation (Safety Population).
Arm/Group | IDP-123 Lotion | Tazorac Cream | Vehicle Lotion | Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/71 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 2/68 | 4/71 | 1/34 | 2/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-123 Lotion (N=68) | Tazorac Cream (N=71) | Vehicle Lotion (N=34) | Vehicle Cream (N=33)
Nasopharyngitis (Infections and infestations) | 2 | 4 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.